CLINICAL TRIAL: NCT01861054
Title: A Single Arm, Preoperative, Pilot Study to Evaluate the Safety and Biological Effects of Orally Administered Reparixin in Early Breast Cancer Patients Who Are Candidates for Surgery
Brief Title: Pilot Study to Evaluate Safety & Biological Effects of Orally Administered Reparixin in Early Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment target not reached
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP0210
Record Dates: First submitted 2013-04-18; First posted 2013-05-23 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: Cancer Stem Cells; Novel targeted therapy; CXCR1/2 Inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — reparixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated patients - Total (Experimental): Patients eligible will be treated with Reparixin as add-in monotherapy
  Interventions: Drug: Reparixin

INTERVENTIONS:
Drug: Reparixin — 1000 mg Oral Reparixin t.i.d. for 21 consecutive days prior to surgery
  Other Names: REP

SUMMARY:
This is a pilot "window of opportunity" clinical study in patients with operable breast cancer investigating use of reparixin as single agent in the time period between clinical diagnosis and surgery.

The primary objectives of this study were:

1- to evaluate the effects of orally administered reparixin on CSCs in the primary tumor and the tumoral microenvironment in an early breast cancer population:

A. CSC were measured in tissue samples by techniques that could include: ALDEFLUOR assay and assessment of CD44/CD24 by flow cytometry, or examination of RNA transcripts by RT-PCR, aldehyde dehydrogenase-1, CD44/CD24 and epithelial mesenchymal transition markers (Snail, Twist, Notch) by immunohistochemistry (IHC). CSC were defined as ALDEFLUOR positive (ALDH-1+) and/or CD44 high/CD24 low by flow cytometry or RT-PCR and IHC and by the detection of ALDH-1+ cells with or without epithelial mesenchymal transition (EMT) transcription factor in IHC assays.

B. Serine-threonine protein kinase (AKT), focal adhesion kinase (FAK), phosphatase and tensin homolog (PTEN) and chemokine receptor-1 (CXCR1) levels were measured in tissue samples by IHC.

C. Measurement of markers of inflammation (interleukin-1beta [IL-1β], interleukin-6 [IL-6], interleukin-8 [IL-8], tumor necrosis factor-alpha [TNF-α], granulocyte macrophage colony stimulating factor [GM-CSF], vascular endothelial growth factor [VEGF], basic fibroblast growth factor [b-FGF] and high-sensitivity C-reactive protein [hsCRP]) in plasma, leukocyte subsets (enumerate T subsets, B, and natural killer/natural killer T [NK/NKT] cells) and study polymorphonuclear leukocyte [PMN] biology in peripheral blood samples. D. Measurement of markers of angiogenesis (CD31 staining), tumor-infiltrating leukocytes (CD4, CD8, NK and macrophages), autophagy (P62 and LC3 by IHC), EpCAM and EMT markers (CD326, CD45, Twist1, SNAIL1, SLUG, ZEB1, FOXC2, TG2, Akt2, P13k and CK19 by RT-PCR) and tissue cellularity (residual disease characterization in tumor bed) in tumor tissue samples.

2. To evaluate the safety of oral reparixin administered three times daily (t.i.d.) for 21 consecutive days.

The secondary objective was to define the pharmacokinetic (PK) profile of orally administered reparixin.

DETAILED DESCRIPTION:
According to the cancer stem cell (CSC) model, tumors are organized in a cellular hierarchy maintained by a subpopulation of cells displaying stem cell properties. These properties include self-renewal (which drives tumorigenesis) and differentiation (which generates the tumor bulk and contributes to cellular heterogeneity).

CSCs were first observed in hematological malignancies but have also been identified in solid tumors of breast, prostate, brain, colon and pancreas. CSCs are thought to be resistant to conventional chemotherapies and this may be why relapse occurs in many patients and this might explain the failure to develop therapies that are consistently able to eradicate solid tumors. Although currently available drugs can shrink metastatic tumors, these effects are usually transient and often do not appreciably extend the life of patients. One reason for the failure of these treatments is the acquisition of drug resistance by the cancer cells as they evolve; another possibility is that existing therapies fail to kill CSCs effectively. Existing therapies have been developed largely against the bulk population of tumor cells because they are often identified by their ability to shrink tumors. Because most cancer cells have limited proliferative potential, an ability to shrink a tumor mainly reflects an ability to kill these cells. It seems that normal stem cells from various tissues tend to be more resistant to chemotherapeutics than mature cell types from the same tissues. The reasons for this are not clear, but may relate to high levels of expression of anti-apoptotic proteins or adenosine triphosphate-binding cassette transporters such as the multidrug resistance gene. If the same were true of CSCs, then one would predict that these cells would be more resistant to chemotherapeutics than tumor cells with limited proliferative potential. Even therapies that cause complete regression of tumors might spare enough CSCs to allow re-growth of the tumors. Therapies that are more specifically directed against CSCs might result in much more durable responses and even cures of metastatic tumors.

There are limited data on the impact of treatment tailoring based on CSC detection. Gene profiling of CSCs could lead to identification of therapeutic targets on CSCs (e.g. hormone receptors (HR), human epidermal growth factor receptor-2 [HER-2] expression, epidermal growth factor receptor [EGFR] expression), and could represent tumor biopsy in "real time". Several groups showed frequent discordance of HER-2 status between primary tumor and CSCs, and case reports showed clinical utility for the use of trastuzumab-based therapy based on HER-2 CSCs status. Similarly, the hormonal status of CSCs could be different from that of the primary tumor, which could lead to increase the number of patients suitable for endocrine therapy, but also could explain why endocrine therapy fails in a subset of HR positive (HR+) patients. More specifically, a recent observation from Ginestier et al. demonstrated that over expression of chemokine receptor 1 (CXCR-1) is associated with the aldehyde dehydrogenase positive (ALDH+) cells. In breast carcinomas, the ALDEFLUOR+ phenotype shows partial overlap with the CD44+CD24-Lin-CSC phenotype. Cellular hierarchies have been identified in a series of molecularly characterized breast cancer cell lines and it has been demonstrated that these lines contained ALDEFLUOR+ components that were both tumorigenic and metastatic in NOD/SCID mice. Furthermore, previous observations demonstrated that the addition of recombinant interleukin-8 (IL-8) increased the CSC population as well as increasing its propensity for invasion. Moreover, tissue damage induced by chemotherapeutic agents may induce IL-8 as part of the injury response. This suggests that strategies aimed at interfering with the IL 8/CXCR-1 axis may be able to target CSCs, increasing the efficacy of current therapies. This experimental data provides another therapeutic target in breast cancer.

Reparixin seems to be a good candidate for use in breast cancer patients because of its very acceptable toxicity profile shown in the Phase I and II clinical trials conducted so far, along with its observed activity in vitro against breast cancer cell lines and in vivo in tumor xenografts in mice. A phase 1 study is currently underway to study the effects of reparixin in combination with paclitaxel in metastatic breast cancer.

This small pilot study aims at exploring the effects on breast CSC markers as well as the safety and PK profile of orally administered single agent reparixin in HER-2 negative (HER-2-) early breast cancer patients in the 3 weeks prior to surgery.

The study will be performed in the interval between disease diagnosis and planned surgery and may lead to a minimal delay in surgery. This is balanced by the potential benefits of the study by evaluating CSCs and their prognostic importance as well as obtaining information about the impact of reparixin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female aged > 18 years.
* Patients with operable breast cancer, with measurable tumors of more than 1 cm in diameter, that are not candidates for neoadjuvant therapy.
* Zubrod (Eastern Co-operative Oncology Group [ECOG]) Performance Status (PS) of 0-1.
* No prior treatment by surgery, radiotherapy, hormone therapy e.g. TAMOXIFEN® or RALOXIFEN® for prevention or chemotherapy.
* Scheduled to undergo definitive local surgery for breast cancer.
* Patients must be willing to undergo two mandatory tumor biopsies (pre and post therapy) that are not required for standard care. A sample of tumor tissue removed during surgery will also be collected for analysis.
* Patients must be able to swallow and retain oral medication (intact tablet).
* Able to undergo all screening assessments outlined in the protocol after giving informed consent.
* Adequate organ function (defined by the following parameters):

  1. Serum creatinine < 140 μmol/L or creatinine clearance > 60 mL/min.
  2. Serum hemoglobin > 9 g/dL; absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L.
  3. Serum bilirubin < upper normal limit (UNL).
  4. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ UNL; alkaline phosphatase (ALP) ≤ UNL; albumin within normal limits.
* Documented hormone receptor (ER and progesterone receptor) and HER-2- status.
* No known hepatitis B virus (unless due to immunization), hepatitis C virus, human immune deficiency virus-I and II positive status.

Exclusion Criteria:

* Male.
* Pregnancy or lactation or unwillingness to use two adequate methods of birth control throughout the study and for 30 days after study discontinuation.
* Any other breast cancer types including inflammatory form.
* Prior surgery to the breast area or primary axillary dissection.
* Prior treatment for breast cancer.
* Use of an investigational drug within 30 days preceding the first dose of study medication.
* Any prior or current cancer, except in situ uterine carcinoma or basocellular cutaneous cancer considered as definitively cured.
* Any associated medical condition considered incompatible with the study, e.g. cardiac, renal, medullar, respiratory or hepatic insufficiency.
* Neurological or psychiatric disorders which may influence understanding of study and informed consent procedures.
* Active or uncontrolled infection.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function.
* Hypersensitivity to:

  1. ibuprofen or to more than one non-steroidal anti-inflammatory drug;
  2. medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2016-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Goldstein, MD, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (9):
- United States (9):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, 4350 Shawnee Mission Pkwy, Suite 1500, Mailstop 6004, Fairway, Kansas
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, MMC Medical Park at Eastchester, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Sara Cannon Research Institute, Nashville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein LJ, Mansutti M, Levy C, Chang JC, Henry S, Fernandez-Perez I, Prausova J, Staroslawska E, Viale G, Butler B, McCanna S, Ruffini PA, Wicha MS, Schott AF; fRida Trial Investigators. A randomized, placebo-controlled phase 2 study of paclitaxel in combination with reparixin compared to paclitaxel alone as front-line therapy for metastatic triple-negative breast cancer (fRida). Breast Cancer Res Treat. 2021 Nov;190(2):265-275. doi: 10.1007/s10549-021-06367-5. Epub 2021 Sep 3. PMID 34476645
- [Derived] Goldstein LJ, Perez RP, Yardley D, Han LK, Reuben JM, Gao H, McCanna S, Butler B, Ruffini PA, Liu Y, Rosato RR, Chang JC. A window-of-opportunity trial of the CXCR1/2 inhibitor reparixin in operable HER-2-negative breast cancer. Breast Cancer Res. 2020 Jan 10;22(1):4. doi: 10.1186/s13058-019-1243-8. PMID 31924241
- See also: Goldstein LJ Breast Cancer Research 22:4. doi: 10.1186/s13058-019-1243-8, 2020 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6954543/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruitment: before initiating a study, the Investigator was required to have written and dated approval from the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) for the study protocol, written informed consent form (ICF), consent form updates, subject recruitment procedures (e.g., advertisements), and any other written information to be provided to subjects.
Pre-assignment Details: It was planned to enroll 2 sub-groups of patients into the study, Group A: ER+ and/or PR+/HER-2- and Group B: ER-/PR-/HER-2-, and the sample size of 20 patients per group was chosen. Twenty patients in total were enrolled, 18 in Group A and 2 in Group B. The study was closed prematurely due to slow enrollment in group B. All 20 patients were included in the Safety Population and 6 (30%) were included in the PK population. All 20 patients completed the study.
Groups:
- ER+ and/or PR+/ HER-2 -: Patients of Group A (estrogen receptor positive (ER+) and/or progesterone receptor positive (PR+)/human epidermal growth factor receptor-2 negative (HER-2-)) were given Reparixin 1000 mg (two 500 mg tablets) for 21 consecutive days. Reparixin was administered orally, every six to eight hours t.i.d. preferably with food. However, if the patient was unable to eat, reparixin could still be administered. Reparixin was administered with about 250 mL water and a light meal or snack.
- ER-/PR-/HER-2-: Patients of Group B (estrogen receptor negative (ER-)/progesterone receptor negative (PR-)/HER-2-) were given Reparixin 1000 mg (two 500 mg tablets) for 21 consecutive days. Reparixin was administered orally, every six to eight hours t.i.d. preferably with food. However, if the patient was unable to eat, reparixin could still be administered. Reparixin was administered with about 250 mL water and a light meal or snack.
Period: Overall Study
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Started | 18 | 2
Safety Population | 18 | 2
PK Population | 4 | 2
Completed | 18 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2- | Total
Number analyzed (Participants) | 18 | 2 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 1 | 17
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (8.92) | 56.5 (12.02) | 54.3 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 2 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 12 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 2 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 21 in Markers of Cancer Stem Cells (CSCs) in the Primary Tumor and the Tumoral Microenvironment (ALDH1,CD44/CD24)
Description: CSCs were measured in tissue samples by the following techniques: ALDH-1 by ALDEFLUOR and by immunohistochemistry (IHC); CD44/CD24 by flow cytometry or examination of RNA transcripts by RT-PCR and by immunohistochemistry (IHC); epithelial mesenchymal markers (Snail, Twist, Notch) by immunohistochemistry (IHC).
Time Frame: At day 21
Population: The Safety Population included all enrolled patients who took at least one dose of study drug reparixin. This population was used for primary endpoints and safety analysis
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 18 | 2
percentage of cells
  ALDH+: number analyzed (Participants) | 14 | 2
  ALDH+ | 1.34 (2.737) | -0.40 (1.131)
  CD44+/CD24-: number analyzed (Participants) | 14 | 2
  CD44+/CD24- | -0.57 (5.617) | 0.20 (1.273)
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Comparison on ALDH+ cells by ALDEFLUOR assay; Test type: Other; p = 0.3149, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Comparison on CD44+/CD24- by flow citometry; Test type: Other; p = 0.8148, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups

2. Primary Outcome: Change From Baseline-1 to Day 21-1 in Pathway Markers by IHC
Description: Pathway markers (AKT, FAK, PTEN and CXCR1) were measured in tissue samples at the pre-study (Day -14 to 0) and Day 21 (or within 24 hours of last dose). For the evaluation of the stain extent, the following semi-quantitative score method (0 to 4) was used: 0, no positive cells; 1, 1-25%; 2, 26-50%; 3, 51-75%; and 4, 76-100%. Hence for this scale, the higher the values, the worse is the outcome. For the evaluation of the stain intensity, the following score method (0 to 3) was used: 0, negative; 1, weak; 2, moderate, 3; strong. Also for this scale, the higher the score, the worse the outcome.
  Serine-threonine protein kinase (AKT, also known as protein kinase B, PKB) Focal adhesion kinase (FAK) Chemokine receptor-1 (CXCR1)
Time Frame: Day 21 (or last day of treatment)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 18 | 2
score on a scale
  Stain Phospho-AKT Extent: number analyzed (Participants) | 12 | 1
  Stain Phospho-AKT Extent | 0 [-1 to 2] | 0 [0 to 0]
  Stain Phospho-AKT Intensity: number analyzed (Participants) | 12 | 1
  Stain Phospho-AKT Intensity | 0 [-1 to 1] | 0 [0 to 0]
  Stain AKT Extent: number analyzed (Participants) | 12 | 1
  Stain AKT Extent | 0 [-4 to 1] | 1.0 [1 to 1]
  Stain AKT Intensity: number analyzed (Participants) | 12 | 1
  Stain AKT Intensity | -0.5 [-3 to 2] | 0 [0 to 0]
  Phospho-FAK Extent: number analyzed (Participants) | 11 | 1
  Phospho-FAK Extent | 0 [-1 to 2] | 0 [0 to 0]
  Phospho-FAK Intensity: number analyzed (Participants) | 11 | 1
  Phospho-FAK Intensity | 0 [-1 to 2] | -1.0 [-1 to -1]
  Stain FAK Extent: number analyzed (Participants) | 12 | 1
  Stain FAK Extent | 0 [-2 to 1] | 1.0 [1 to 1]
  Stain FAK Intens: number analyzed (Participants) | 12 | 1
  Stain FAK Intens | 0 [-2 to 2] | 0 [0 to 0]
  Stain C-PTEN Extent: number analyzed (Participants) | 12 | 1
  Stain C-PTEN Extent | 0 [-4 to 2] | 0 [0 to 0]
  Stain C-PTEN Intensity: number analyzed (Participants) | 12 | 1
  Stain C-PTEN Intensity | 0 [-2 to 1] | 0 [0 to 0]
  Stain D-PTEN Extent: number analyzed (Participants) | 12 | 1
  Stain D-PTEN Extent | 0 [-4 to 2] | 0 [0 to 0]
  Stain D-PTEN Intensity: number analyzed (Participants) | 12 | 1
  Stain D-PTEN Intensity | 0 [-2 to 1] | 0 [0 to 0]
  Stain CXCR1 Extent: number analyzed (Participants) | 12 | 1
  Stain CXCR1 Extent | 0 [-4 to 1] | 1.0 [1 to 1]
  Stain CXCR1 Intensity: number analyzed (Participants) | 12 | 1
  Stain CXCR1 Intensity | -0.5 [-3 to 1] | 1.0 [1 to 1]
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Phospho AKT Extent; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Phospho-AKT Intensity; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; AKT Extent; Test type: Other; p = 0.2245, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; AKT Intensity; Test type: Other; p = 0.5785, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Phospho-FAK Extent; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Phospho-FAK Intensity; Test type: Other; p = 0.3139, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; FAK Extent; Test type: Other; p = 0.2120, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; FAK Intensity; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; C-PTEN Extent; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; C-PTEN Intensity; Test type: Other; p = 0.8728, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; D-PTEN Extent; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; D-PTEN Intensity; Test type: Other; p = 0.8728, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CXCR1 Extent; Test type: Other; p = 0.2265, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CXCR1 Intensity; Test type: Other; p = 0.2403, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change From Baseline to Day 21 in Markers of Inflammation
Description: Markers of inflammation (IL-1β, IL-6, IL-8, TNF-α, GM-CSF, VEGF, and b-FGF) were measured in plasma from peripheral blood.
  IL = interleukins TNF-α = tumor necrosis factor-alpha GM-CSF = macrophage colony stimulating factor VEGF = vascular endothelial growth factor b-FGF = basic fibroblast growth factor
Time Frame: At Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ML
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 18 | 2
pg/ML
  Interleukin 1 Beta: number analyzed (Participants) | 16 | 2
  Interleukin 1 Beta | 7.019 (30.3118) | 0 (0.000)
  Interleukin 6: number analyzed (Participants) | 16 | 2
  Interleukin 6 | 9.593 (39.2733) | 0 (0)
  Interleukin 8: number analyzed (Participants) | 16 | 2
  Interleukin 8 | -25.874 (134.3213) | 29.320 (41.6910)
  TNFα: number analyzed (Participants) | 16 | 2
  TNFα | 2.669 (8.0313) | -0.890 (3.5780)
  GM-CSF: number analyzed (Participants) | 16 | 2
  GM-CSF | -2.678 (8.2154) | 8.705 (12.3107)
  VEGF: number analyzed (Participants) | 16 | 2
  VEGF | 253.584 (1120.6125) | 27.635 (39.0818)
  b-FGF: number analyzed (Participants) | 16 | 2
  b-FGF | 20.164 (93.4614) | -9.750 (13.7886)
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Interleukin 1 Beta; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Interleukin 6; Test type: Other; p = 0.6945, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 3: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Interleukin 8; Test type: Other; p = 0.9448, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 4: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Tumor Necrosis Factor - alpha; Test type: Other; p = 0.6292, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 5: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Granulocyte Macrophage Colony Stm Factor; Test type: Other; p = 0.2354, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 6: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Vascular Endothelial Growth Factor; Test type: Other; p > 0.9999, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 7: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Basic Fibroblast Growth Factor; Test type: Other; p = 0.4719, Wilcoxon (Mann-Whitney) — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups

4. Primary Outcome: Change From Baseline-1 to Day 21-1 in Markers of Angiogenesis (CD31 Staining)
Description: CD31 staining by IHC. For the evaluation of the stain extent, the following semi-quantitative score method (0 to 4) was used: 0, no positive cells; 1, 1-25%; 2, 26-50%; 3, 51-75%; and 4, 76-100%. Hence for this scale, the higher the values, the worse is the outcome. For the evaluation of the stain intensity, the following score method (0 to 3) was used: 0, negative; 1, weak; 2, moderate, 3; strong. Also for this scale, the higher the score, the worse the outcome.
  CD31 is a transmembrane glycoprotein, 130-140 kDa, also know as platelet-endothelium cell adhesion molecule (PECAM-1). CD31 is ligand for CD38 and plays a role in thrombosis and angiogenesis. CD31 is strongly expressed in endothelial cells and weakly expressed in megakaryocytes, platelets, occasional plasma cells, lymphocytes (espc. marginal zone B-cells, peripheral T-cells) and neutrophils.
Time Frame: At day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 18 | 2
score on a scale
  Stain CD31 Extent: number analyzed (Participants) | 12 | 1
  Stain CD31 Extent | 0 [-2 to 1] | 1.0 [1 to 1]
  Stain CD31 Intensity: number analyzed (Participants) | 12 | 1
  Stain CD31 Intensity | 0 [-1 to 1] | 1.0 [1 to 1]
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD31 Extent; Test type: Other; p = 0.0951, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD31 Intensity; Test type: Other; p = 0.1643, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change From Baseline-1 to Day 21-1 in Markers of Autophagy (P62 and LC3B by IHC)
Description: Autophagy is a lysosomal degradation and recycling process implicated in cancer progression and therapy resistance. Labeling of p62 serves as a useful marker for the induction of autophagy, clearance of protein aggregates, and the inhibition of autophagy. Labeling of LC3B serves to track the binding of p62 and subsequent recruitment of autophagosomes.
  For the evaluation of the extent, the following semi-quantitative score method (0 to 4) was used: 0, no positive cells; 1, 1-25%; 2, 26-50%; 3, 51-75%; and 4, 76-100%. Hence for this scale, the higher the values, the worse is the outcome. For the evaluation of the intensity, the following score method (0 to 3) was used: 0, negative; 1, weak; 2, moderate, 3; strong. Also for this scale, the higher the score, the worse the outcome.
Time Frame: At day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 18 | 2
score on a scale
  Stain P62 Extent: number analyzed (Participants) | 12 | 1
  Stain P62 Extent | -1.0 [-3 to 1] | 0 [0 to 0]
  Stain P62 Intensity: number analyzed (Participants) | 12 | 1
  Stain P62 Intensity | 0 [-2 to 0] | -1.0 [-1 to -1]
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; P62 Extent; Test type: Other; p = 0.4183, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; P62 Intensity; Test type: Other; p = 0.3702, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Pharmacokinetics of Reparixin (DF1681Y, DF1681Y Unbound, DF2243Y, DF2188Y) - Cmax
Description: Once absorbed, reparixin is highly protein bound. By comparing Cmax and AUC for unbound drug to that for total drug, only < 0.1% to 0.2% of reparixin is available as unbound (free) drug. The intent of the PK outcomes was not to compare the results between the two cohorts; for this reason results for the PK outcomes are reported for the whole group of the treated patients.
  Cmax = Maximum plasma concentration obtained directly from the data without interpolation, expressed in concentration units
Time Frame: At Days 1 (pre-first dose and 0.25, 0.5, 1, 2, 4, 6, 8h post dose) and 21(pre-first dose and 0.25, 0.5, 1, 2, 4, 6, 8h post dose)
Population: The PK Population consisted of patients who received at least one dose of reparixin and had at least one valid, quantifiable PK parameter. This population was used for PK analyses.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Groups:
- Treated Patients - Total: Patients eligible were treated with Reparixin as add-in monotherapy
  Reparixin: 1000 mg Oral Reparixin t.i.d. for 21 consecutive days prior to surgery
Arm/Group | Treated Patients - Total
Number analyzed (Participants) | 6
micrograms/mL
  Day1 - DF1681Y | 62.925 (31.5024)
  Day21 - DF1681Y | 63.927 (15.7616)
  Day1 - DF1681Y unbound | 145.167 (116.6114)
  Day21 - DF1681Y unbound | 136.552 (104.8681)
  Day 1 - DF2243Y | 15.788 (2.5240)
  Day 21 - DF2243Y | 20.812 (9.9776)
  Day 1 - DF2188Y | 7.302 (1.5129)
  Day 21 - DF2188Y | 10.367 (4.3439)

7. Secondary Outcome: Pharmacokinetics of Reparixin (DF1681Y, DF1681Y Unbound, DF2243Y, DF2188Y) - Tmax and T1/2
Description: Once absorbed, reparixin is highly protein-bound. By comparing Cmax and AUC for unbound drug to that for total drug, only < 0.1% to 0.2% of reparixin is available as unbound (free) drug. The intent of the PK outcomes was not to compare the results between the two cohorts; for this reason results for the PK outcomes are reported for the whole group of the treated patients.
  tmax = Time to reach the maximum plasma concentration obtained directly from the data without interpolation t1/2 = Terminal elimination half-life calculated as ln(2)/ lambda z; calculated only if the coefficient of determination R2 in lambda z estimation is at least 0.8.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treated Patients - Total
Number analyzed (Participants) | 6
hours
  Day1 - DF1681Y tmax | 2.667 (2.8752)
  Day21 - DF1681Y tmax | 0.997 (0.5508)
  Day1 - DF1681Y unbound tmax | 1.583 (1.2813)
  Day21 - DF1681Y unbound tmax | 1.092 (0.4903)
  Day 1 - DF2243Y tmax | 4.333 (2.3381)
  Day 21 - DF2243Y tmax | 2.331 (0.8179)
  Day 1 - DF2188Y tmax | 2.500 (1.2247)
  Day 21 - DF2188Y tmax | 1.508 (0.5389)
  Day1 - DF1681Y t1/2: number analyzed (Participants) | 4
  Day1 - DF1681Y t1/2 | 2.090 (0.9847)
  Day21 - DF1681Y t1/2 | 1.626 (0.4068)
  Day1 - DF1681Y unbound t1/2: number analyzed (Participants) | 3
  Day1 - DF1681Y unbound t1/2 | 1.403 (0.4592)
  Day21 - DF1681Y unbound t1/2 | 0.989 (0.1683)
  Day 1 - DF2243Y t1/2: number analyzed (Participants) | 2
  Day 1 - DF2243Y t1/2 | 1.913 (0.3268)
  Day 21 - DF2243Y t1/2: number analyzed (Participants) | 4
  Day 21 - DF2243Y t1/2 | 2.575 (0.6442)
  Day 1 - DF2188Y t1/2: number analyzed (Participants) | 4
  Day 1 - DF2188Y t1/2 | 2.035 (1.0618)
  Day 21 - DF2188Y t1/2: number analyzed (Participants) | 5
  Day 21 - DF2188Y t1/2 | 1.575 (0.1953)

8. Secondary Outcome: Pharmacokinetics of Reparixin (DF1681Y, DF1681Y Unbound, DF2243Y, DF2188Y) - AUC0-8, AUCinf, AUClast, AUCtau at Day 21,
Description: The intent of the PK outcomes was not to compare the results between the two cohorts; for this reason results for the PK outcomes are reported for the whole group of the treated patients.
  AUC0-8 = The area under the plasma concentration-time curve from time 0 to 8 hours post-dose; AUClast = The area under the concentration-time curve from time 0 to last quantifiable concentration AUCtau = The area under the plasma concentration-time curve for dosing interval (dosing interval [tau] = 8 hours); AUCinf = The total area under the plasma concentration-time curve from time zero to time infinity; AUC0-inf = AUClast + Clast/lambda zeta, where Clast is the last observed concentration ≥ lower limit of quantitation at time tlast.
  All these parameters were calculated by the linear trapezoidal rule.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Treated Patients - Total
Number analyzed (Participants) | 6
h*μg/mL
  DF1681Y - AUC0-8 - Day 1 | 189.357 (60.2362)
  DF1681Y - AUC0-8 - Day 21 | 174.303 (29.8012)
  DF1681Y unbound- AUC0-8 - Day 1 | 222.602 (128.0328)
  DF1681Y unbound- AUC0-8 - Day 21 | 233.382 (166.0402)
  DF2243Y - AUC0-8 - Day 1: number analyzed (Participants) | 5
  DF2243Y - AUC0-8 - Day 1 | 78.469 (18.8116)
  DF2243Y - AUC0-8 - Day 21: number analyzed (Participants) | 4
  DF2243Y - AUC0-8 - Day 21 | 105.001 (58.2634)
  DF2188Y - AUC0-8 - Day 1 | 31.040 (7.9369)
  DF2188Y - AUC0-8 - Day 21: number analyzed (Participants) | 5
  DF2188Y - AUC0-8 - Day 21 | 33.395 (13.2129)
  DF1681Y - AUCinf - Day 1: number analyzed (Participants) | 4
  DF1681Y - AUCinf - Day 1 | 211.243 (71.4823)
  DF1681Y - AUCinf - Day 21 | 182.479 (36.1551)
  DF1681Y unbound - AUCinf - Day 1: number analyzed (Participants) | 3
  DF1681Y unbound - AUCinf - Day 1 | 235.152 (180.1547)
  DF1681Y unbound - AUCinf - Day 21 | 234.547 (166.3017)
  DF2243Y - AUCinf - Day 1: number analyzed (Participants) | 2
  DF2243Y - AUCinf - Day 1 | 71.297 (25.6857)
  DF2243Y - AUCinf - Day 21: number analyzed (Participants) | 4
  DF2243Y - AUCinf - Day 21 | 129.275 (74.5406)
  DF2188Y - AUCinf - Day 1: number analyzed (Participants) | 4
  DF2188Y - AUCinf - Day 1 | 31.669 (11.2792)
  DF2188Y - AUCinf - Day 21: number analyzed (Participants) | 5
  DF2188Y - AUCinf - Day 21 | 35.092 (13.9473)
  DF1681Y - AUClast - Day 1 | 189.319 (60.2817)
  DF1681Y - AUClast - Day 21 | 172.296 (28.1847)
  DF1681Y unbound - AUClast - Day 1 | 222.078 (128.1305)
  DF1681Y unbound - AUClast - Day 21 | 231.235 (167.0377)
  DF2243Y - AUClast - Day 1 | 76.821 (17.3033)
  DF2243Y - AUClast - Day 21 | 97.360 (46.6809)
  DF2188Y - AUClast - Day 1 | 31.028 (7.9336)
  DF2188Y - AUClast - Day 21 | 35.433 (12.8434)
  DF1681Y - AUCtau - Day 21 | 174.303 (29.8012)
  DF1681Y unbound - AUCtau - Day 21 | 233.382 (166.0402)
  DF2243Y - AUCtau - Day 21: number analyzed (Participants) | 4
  DF2243Y - AUCtau - Day 21 | 105.001 (58.2634)
  DF2188Y - AUCtau - Day 21: number analyzed (Participants) | 5
  DF2188Y - AUCtau - Day 21 | 33.395 (13.2129)

9. Secondary Outcome: Pharmacokinetics of Reparixin (DF1681Y, DF1681Y Unbound, DF2243Y, DF2188Y) - CL/F (L/h) at Day 1, CLSS/F (L/h) Day 21)
Description: The intent of the PK outcomes was not to compare the results between the two cohorts; for this reason results for the PK outcomes are reported for the whole group of the treated patients.
  CL/F = Apparent oral clearance - for DF1681Y only, calculated as dose/AUCinf.; calculated only when the coefficient of determination R2 in lambda zeta estimation is at least 0.8 and percent AUC extrapolation is less than or equal to 20%.
  CLss/F = Steady state apparent oral clearance - for DF1681Y only calculated as dose/AUCtau.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Treated Patients - Total
Number analyzed (Participants) | 6
L/h
  DF1681Y - CL/F - Day 1: number analyzed (Participants) | 4
  DF1681Y - CL/F - Day 1 | 5.173 (1.7466)
  DF1681Y - CLSS/F - Day 21 | 5.866 (0.9086)
  DF1681Y unbound - CL/F - Day 1: number analyzed (Participants) | 3
  DF1681Y unbound - CL/F - Day 1 | 7156.189 (6334.8463)
  DF1681Y unbound - CLSS/F - Day 21 | 5604.781 (2335.8016)

10. Secondary Outcome: Change From Baseline to Day 21 in Leukocytes Subsets
Description: The Leukocytes subsets analyzed are the following: Lymphocyte in WBC, Total T cell in lymphocytes, B cells in lymphocytes, T-helper cell in lymphocytes, CTL in lymphocytes, NKT cell in lymphocytes, ADCC NK subsets in lymphocytes, Regulatory NK subsets in lymphocytes, Exhausted NK subsets in lymphocytes, CD56-CD16+ NK subsets in lymphocytes, CD11b in PMNs - IL-8, CD18 in PMNs - IL-8, MFI of CD11b - IL-8, MFI of CD66b - IL-8, MFI of CD18 - IL-8, CD11b in PMNs - US, CD18 in PMNs - US, MFI of CD11b - US, MFI of CD66b - US, MFI of CD18 - US, Percent Monocytes expressing IL6 - IL-8,Percent Monocytes expressing IL1b - IL-8, Percent Monocytes expressing IL8 - IL-8, Percent Monocytes expressing TNFa - IL-8, Percent Neutrophils expressing IL6 - IL-8, Percent Neutrophils expressing IL1b - IL-8, Percent Neutrophils expressing IL8 - IL-8, Percent Neutrophils expressing TNFa - IL-8,Percent Monocytes expressing IL6 - US,Percent Monocytes expressing IL1b - US, etc.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of total
Arm/Group | ER+ and/or PR+/ HER-2 - | ER-/PR-/HER-2-
Number analyzed (Participants) | 16 | 1
percent of total
  Lymphocyte in WBC | -2.51 (9.099) | -3.70 (NA) — Since the patient is only one, no SD can be calculated
  Total T cell in lymphocytes | 1.28 (4.602) | -2.80 (NA) — Since the patient is only one, no SD can be calculated
  B cell in lymphocytes | 2.678 (7.5565) | 43.190 (NA) — Since the patient is only one, no SD can be calculated
  T-helper cell in lymphocytes | -1.44 (5.158) | -24.90 (NA) — Since the patient is only one, no SD can be calculated
  CTL in lymphocytes | -0.639 (5.5106) | -24.100 (NA) — Since the patient is only one, no SD can be calculated
  NKT cell in lymphocytes | 0.510 (1.5759) | 0.140 (NA) — Since the patient is only one, no SD can be calculated
  ADCC NK subsets in lymphocytes | 0.727 (4.1787) | 1.430 (NA) — Since the patient is only one, no SD can be calculated
  Regulatory NK subsets in lymphocytes | -1.358 (3.2465) | 0.370 (NA) — Since the patient is only one, no SD can be calculated
  Exhausted NK subsets in lymphocytes | -0.177 (1.7006) | -0.170 (NA) — Since the patient is only one, no SD can be calculated
  CD56-CD16+ NK subsets in lymphocytes | 0.708 (1.6772) | 0.310 (NA) — Since the patient is only one, no SD can be calculated
  CD11b in PMNs - IL-8 | -1.48 (4.877) | -11.60 (NA) — Since the patient is only one, no SD can be calculated
  CD18 in PMNs - IL-8 | -0.23 (4.104) | 2.10 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD11b - IL-8 | -1.63 (2.205) | 3.50 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD66b - IL-8 | -3.9 (507.79) | -929.0 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD18 - IL-8 | -13.0 (495.89) | 71.0 (NA) — Since the patient is only one, no SD can be calculated
  CD11b in PMNs - US | 1.56 (9.515) | -4.20 (NA) — Since the patient is only one, no SD can be calculated
  CD18 in PMNs - US | -5.758 (23.7696) | -0.400 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD11b - US | -0.84 (1.571) | -0.30 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD66b - US | 35.1 (536.54) | -757.0 (NA) — Since the patient is only one, no SD can be calculated
  MFI of CD18 - US | -105.64 (679.547) | -47.00 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL6 - IL-8: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL6 - IL-8 | 8.40590 (27.654326) | 0.52600 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL1b - IL-8: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL1b - IL-8 | 8.27479 (24.364503) | 0.32600 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL8 - IL-8: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL8 - IL-8 | -0.35947 (3.983235) | -0.04400 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing TNFa - IL-8: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing TNFa - IL-8 | 0.40504 (1.906309) | -0.39900 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL6 - IL-8: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL6 - IL-8 | 2.83019 (26.145843) | 0.36340 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL1b - IL-8: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL1b - IL-8 | 10.24530 (32.068081) | 0.33400 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL8 - IL-8: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL8 - IL-8 | 0.04596 (1.667000) | 0.05742 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing TNFa - IL-8: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing TNFa - IL-8 | 0.35635 (2.269023) | 0.03500 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL6 - US: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL6 - US | 9.77675 (29.705447) | 0.26500 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL1b - US: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL1b - US | 5.58031 (28.862940) | 1.03400 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL8 - US: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing IL8 - US | 0.14087 (2.716051) | -0.27600 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing TNFa - US: number analyzed (Participants) | 15 | 1
  Percent Monocytes expressing TNFa - US | -0.11532 (1.333406) | 0.28200 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL6 - US: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL6 - US | 5.50297 (21.932274) | 0.59260 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL1b - US: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL1b - US | 9.28329 (33.754437) | 1.36450 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL8 - US: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing IL8 - US | 0.45567 (2.053990) | 0.15020 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing TNFa - US: number analyzed (Participants) | 15 | 1
  Percent Neutrophils expressing TNFa - US | 0.46929 (2.876200) | 0.54910 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL6 - LPS: number analyzed (Participants) | 14 | 1
  Percent Monocytes expressing IL6 - LPS | -0.23 (8.015) | -9.60 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL1b - LPS: number analyzed (Participants) | 14 | 1
  Percent Monocytes expressing IL1b - LPS | -5.18 (18.237) | 27.80 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL8 - LPS: number analyzed (Participants) | 14 | 1
  Percent Monocytes expressing IL8 - LPS | -4.2057 (21.72201) | -74.3700 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing TNFa - LPS: number analyzed (Participants) | 14 | 1
  Percent Monocytes expressing TNFa - LPS | -3.145 (8.8075) | -56.400 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL6 - LPS: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL6 - LPS | -2.0310 (4.60857) | 72.3690 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL1b - LPS: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL1b - LPS | -1.68086 (5.470114) | 78.19200 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL8 - LPS: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL8 - LPS | 0.14986 (1.844687) | 1.18700 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing TNFa - LPS: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing TNFa - LPS | 0.1497 (1.97537) | 1.7720 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL6 - LPS+IL-8: number analyzed (Participants) | 13 | 1
  Percent Monocytes expressing IL6 - LPS+IL-8 | -3.42 (6.783) | 1.20 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL1b - LPS+IL-8: number analyzed (Participants) | 13 | 1
  Percent Monocytes expressing IL1b - LPS+IL-8 | -4.79 (14.168) | 25.90 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing IL8 - LPS+IL-8: number analyzed (Participants) | 13 | 1
  Percent Monocytes expressing IL8 - LPS+IL-8 | -7.738 (12.9421) | -76.990 (NA) — Since the patient is only one, no SD can be calculated
  Percent Monocytes expressing TNFa - LPS+IL-8: number analyzed (Participants) | 13 | 1
  Percent Monocytes expressing TNFa - LPS+IL-8 | -0.3018 (9.97119) | -57.9100 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL6 - LPS+IL-8: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL6 - LPS+IL-8 | 1.2629 (20.77484) | 62.7900 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL1b - LPS+IL-8: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL1b - LPS+IL-8 | 0.1980 (27.96300) | 81.6290 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing IL8 - LPS+IL-8: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing IL8 - LPS+IL-8 | 0.0348 (1.81583) | 1.0010 (NA) — Since the patient is only one, no SD can be calculated
  Percent Neutrophils expressing TNFa - LPS+IL-8: number analyzed (Participants) | 14 | 1
  Percent Neutrophils expressing TNFa - LPS+IL-8 | -0.0349 (1.75308) | 2.6490 (NA) — Since the patient is only one, no SD can be calculated
  Percent FITC eColi Control: number analyzed (Participants) | 13 | 1
  Percent FITC eColi Control | 4.327 (7.7795) | -8.500 (NA) — Since the patient is only one, no SD can be calculated
  Percent FITC eColi Test: number analyzed (Participants) | 13 | 1
  Percent FITC eColi Test | -1.056 (3.6456) | -4.200 (NA) — Since the patient is only one, no SD can be calculated
  Percent PMNs unstimulated: number analyzed (Participants) | 13 | 1
  Percent PMNs unstimulated | -5.025 (16.3554) | 28.690 (NA) — Since the patient is only one, no SD can be calculated
  Percent PMNs fMLP: number analyzed (Participants) | 13 | 1
  Percent PMNs fMLP | 9.152 (18.2092) | 23.300 (NA) — Since the patient is only one, no SD can be calculated
  Percent L-selectin unstimulated: number analyzed (Participants) | 13 | 1
  Percent L-selectin unstimulated | 4.341 (25.8071) | -25.000 (NA) — Since the patient is only one, no SD can be calculated
  Percent L-selectin fMLP: number analyzed (Participants) | 13 | 1
  Percent L-selectin fMLP | -0.2845 (0.95877) | -0.2460 (NA) — Since the patient is only one, no SD can be calculated
Statistical Analysis 1: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Lymphocyte in WBC; Test type: Other; p = 0.6168, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 2: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Total T cell in lymphocytes; Test type: Other; p = 0.6168, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 3: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; B cell in lymphocytes; Test type: Other; p = 0.1453, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 4: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; T-helper cell in lymphocytes; Test type: Other; p = 0.1453, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 5: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CTL in lymphocytes; Test type: Other; p = 0.1453, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 6: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; NKT cell in lymphocytes; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 7: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; ADCC NK subsets in lymphocytes; Test type: Other; p = 0.7634, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 8: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Regulatory NK subsets in lymphocytes; Test type: Other; p = 0.5487, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 9: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Exhausted NK subsets in lymphocytes; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 10: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD56-CD16+ NK subsets in lymphocytes; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 11: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD11b in PMNs - IL-8; Test type: Other; p = 0.1451, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 12: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD18 in PMNs - IL-8; Test type: Other; p = 0.2779, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 13: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD11b - IL-8; Test type: Other; p = 0.1444, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 14: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD66b - IL-8; Test type: Other; p = 0.1453, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 15: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD18 - IL-8; Test type: Other; p = 0.9200, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 16: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD11b in PMNs - US; Test type: Other; p = 0.2779, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 17: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; CD18 in PMNs - US; Test type: Other; p = 0.6164, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 18: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD11b - US; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 19: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD66b - US; Test type: Other; p = 0.2032, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 20: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; MFI of CD18 - US; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 21: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL6 - IL-8; Test type: Other; p = 0.5250, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 22: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL1b - IL-8; Test type: Other; p = 0.6706, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 23: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL8 - IL-8; Test type: Other; p = 0.8312, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 24: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing TNFa - IL-8; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 25: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL6 - IL-8; Test type: Other; p = 0.2952, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 26: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL1b - IL-8; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 27: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL8 - IL-8; Test type: Other; p = 0.2952, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 28: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing TNFa - IL-8; Test type: Other; p = 0.5250, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 29: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL6 - US; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 30: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL1b - US; Test type: Other; p = 0.2952, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 31: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL8 - US; Test type: Other; p > 0.9999, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 32: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing TNFa - US; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 33: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL6 - US; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 34: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL1b - US; Test type: Other; p = 0.2952, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 35: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL8 - US; Test type: Other; p = 0.3992, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 36: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing TNFa - US; Test type: Other; p = 0.2952, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 37: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL6 - LPS; Test type: Other; p = 0.2238, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 38: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL1b - LPS; Test type: Other; p = 0.2238, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 39: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL8 - LPS; Test type: Other; p = 0.1543, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 40: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing TNFa - LPS; Test type: Other; p = 0.1547, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 41: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL6 - LPS; Test type: Other; p = 0.1547, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 42: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL1b - LPS; Test type: Other; p = 0.1547, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 43: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL8 - LPS; Test type: Other; p = 0.4314, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 44: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing TNFa - LPS; Test type: Other; p = 0.3153, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 45: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL6 - LPS+IL-8; Test type: Other; p = 0.4700, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 46: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL1b - LPS+IL-8; Test type: Other; p = 0.1605, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 47: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing IL8 - LPS+IL-8; Test type: Other; p = 0.1605, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 48: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Monocytes expressing TNFa - LPS+IL-8; Test type: Other; p = 0.1605, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 49: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL6 - LPS+IL-8; Test type: Other; p = 0.1547, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 50: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL1b - LPS+IL-8; Test type: Other; p = 0.1547, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 51: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing IL8 - LPS+IL-8; Test type: Other; p = 0.3153, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 52: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent Neutrophils expressing TNFa - LPS+IL-8; Test type: Other; p = 0.1543, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 53: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent FITC eColi Control; Test type: Other; p = 0.1601, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 54: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent FITC eColi Test; Test type: Other; p = 0.2368, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 55: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent PMNs unstimulated; Test type: Other; p = 0.1605, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 56: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent PMNs fMLP; Test type: Other; p = 0.4700, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 57: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent L-selectin unstimulated; Test type: Other; p = 0.3392, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups
Statistical Analysis 58: Comparison: ER+ and/or PR+/ HER-2 - vs ER-/PR-/HER-2-; Percent L-selectin fMLP; Test type: Other; p = 0.8080, t-test, 2 sided — P-Value is based on two-sample t-test or Wilcoxon Rank-Sum test, where appropriate, comparing the 2 study groups

ADVERSE EVENTS:
Time Frame: throughout the study and at OTV (off treatment visit) up to the 30 days after the last dose of reparixin
Groups:
- Total: This represents the total safety population of 20 patients
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=20)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=20)
Nausea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 8
Pain (General disorders) | 2
Oedema peripheral (General disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 5
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Pheripheral sensory neuropathy (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Insomnia (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 1
Mood swings (Psychiatric disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Eye infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Epidermolysis (Congenital, familial and genetic disorders) | 1
Vision blurred (Eye disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No